CLINICAL TRIAL: NCT07406750
Title: Hemodynamic Diagnostic Ultrasound of Venous Congestion (VExUS) Performed by Intensive Care Nurses on Patients With Sepsis.
Brief Title: Hemodynamic Venous Congestion Ultrasound (VExUS) by ICU Nurses in Sepsis Patients.
Acronym: VEXIVAN
Status: Not yet recruiting | Type: Observational
Sponsor: Region Örebro County (Other)
Collaborators: Örebro University, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: JS009
Record Dates: First submitted 2025-11-25; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Sepsis; Sepsis and Septic Shock; Sepsis at Intensive Care Unit; Intensive Care Nurses
Keywords: sepsis; intensive care; ultrasound; venous congestion; VExUS; intensive care nurse
MeSH Terms: conditions — Sepsis; Shock, Septic; Hyperemia | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive care nurse: Intensive care nurses that perform hemodynamic diagnostic ultrasound acording to the VExUS protocol
  Interventions: Behavioral: Education in performing hemodynamic diagnostic ultrasound of venous congestion
- Intensive care patients: Intensive care patients with sepsis
  Interventions: Diagnostic Test: Hemodynamic diagnostic ultrasound of venous congestion

INTERVENTIONS:
Behavioral: Education in performing hemodynamic diagnostic ultrasound of venous congestion — Educational program in performing hemodynamic diagnostic ultrasound of venous congestion
  Groups: Intensive care nurse
Diagnostic Test: Hemodynamic diagnostic ultrasound of venous congestion — Hemodynamic diagnostic ultrasound of venous congestion
  Other Names: VeXUS
  Groups: Intensive care patients

SUMMARY:
Sepsis is a serious condition where the body's immune response to infection overreacts, leading to organ damage and death. Venous congestion, a buildup of blood in the veins, can occur in sepsis and contribute to organ injury. VExUS (Venous Excess Ultrasound Score) is an ultrasound method that can detect congestion early. This study examines whether ICU nurses, after training, can perform VExUS reliably, explores their experiences, and investigates links between VExUS findings and clinical outcomes.

DETAILED DESCRIPTION:
Sepsis is a serious and potentially life-threatening condition that happens when the body's defense system overreacts to an infection. This overreaction can reduce the oxygen supply to the body's organs, causing damage and, in severe cases, organ failure. Up to 30% of people with sepsis die from it, and it is one of the most common causes of death in intensive care units.

Venous congestion, which means blood builds up in the veins, can occur in sepsis-for example, due to fluid overload or reduced heart function. This condition has been linked to organ injury. The VExUS (Venous Excess Ultrasound Score) is an ultrasound-based method that evaluates blood flow in the body's main veins. It has shown promise for identifying patients with venous congestion early. By using VExUS, it may be possible to detect the risk of organ injury sooner in intensive care patients with sepsis.

Ultrasound is becoming an increasingly important diagnostic tool in intensive care and is now often used directly at the bedside. Doctors already use ultrasound in many clinical situations and have extensive experience with it. Intensive care nurses, however, have had less opportunity to use ultrasound. Increasing their skills in this area could improve patient care.

VExUS is a relatively simple method that assesses blood flow in central veins without requiring precise measurements, making it well suited as an introduction to ultrasound use.

The purpose of this study is to examine whether intensive care nurses, after training, can perform VExUS on sepsis patients reliably. In the long term, this study could lead to intensive care nurses routinely performing VExUS as part of their hemodynamic assessment of patients.The study also explores the nurses' experiences and confidence with the method, including interviews. In addition, it investigates whether venous congestion identified by VExUS is linked to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Intensive Care Nurses a) Intensive care nurse, specialist degree in intensive care. b) ≥1,5 years of experience in intensive care. c) ≥75% clinical employment rate at the ICU. d) Continued employment until 2026 at the ICU at Örebro University Hospital. e) Written informed consent Intensive Care Patients

1. Patients with suspected or verified sepsis according to the Sepsis 3 criteria (suspected or confirmed infection), ≥qSOFA (systolic blood pressure < 90 mmHg, GCS ≤ 13, respiratory rate ≥ 22 per minute) or rise in SOFA score ≥ 2 points and admitted to the ICU.
2. ≥18 years of age.

Exclusion Criteria:

Intensive Care Nurses

a) Personnel with primarily an administration position or less clinical duty at the ICU.

Intensive Care Patients

1. Patients with preexisting liver cirrhosis.
2. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intensive care nurses with a specialist degree in intensive care and intensive care patients with sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Intensive care nurses' VExUS performance | two years
  Intensive care nurses' performance, regarding ultrasound image quality and assessment of ultrasound images according to VExUS protocol, evaluated by two experts.

SECONDARY OUTCOMES:
Intra-rater VExUS reliability | two years
  Agreement of assessments of prior collected ultrasound images, according to VExUS protocol, performed by the same intensive care nurse.
Inter-rater VExUS reliability | two years
  Agreement of assessments of prior collected ultrasound images according to VExUS protocol performed by different intensive care nurses.
Inter-rater VExUS image agreement | two years
  Agreement of the ability to obtain ultrasound images according to VExUS protocol performed on the same intensive care patients by different intensive care nurses, in temporal proximity.
Venous congestion measured by VExUS and fluid status | two years
  Association of presence of venous congestion assessed by VExUS over time in septic intensive care patients and daily measures used to monitor fluid status, such as daily weight, daily fluid balance and cumulative fluid balance.
Venous congestion measured by VExUS and clinical outcomes | two years
  Association of presence of venous congestion assessed by VExUS over time in septic intensive care patients and clinical outcomes determined by mortality in the ICU, 30 days mortality, ICU length of stay, hospital length of stay, SOFA score, time in assisted ventilation, need of vasoactive agents, gastrointestinal dysfunction, acute kidney injury and physiological variables.
Intensive care nurses' self-efficacy, confidence and experiences | two years
  Differences in intensive care nurses' perceived self-efficacy and confidence at various time points during data collection, along with their experiences.

IPD SHARING:
Plan to Share IPD: No